CLINICAL TRIAL: NCT00063778
Title: A Phase I Safety and Immunogenicity Trial of an Alphavirus Replicon HIV Subtype C Gag Vaccine (AVX101, Alphavax, Inc.) in Healthy HIV-1 Uninfected Adult Volunteers
Brief Title: Safety of an HIV Vaccine (AVX101) in HIV Uninfected Volunteers in the United States and South Africa
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AlphaVax, Inc. (Industry)
Collaborators: HIV Vaccine Trials Network (Network); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HVTN 040
Record Dates: First submitted 2003-07-07; First posted 2003-07-08 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV Preventive Vaccine; AIDS Vaccines; Gene Products, gag; HIV-1; Dose-Response Relationship, Immunologic; Injections, Subcutaneous
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 x 10^4 IU dose (Experimental): Vaccine dose of 1 x 10^4 IU per injection
  Interventions: Biological: AVX101
- 1 x 10^5 IU dose (Experimental): Vaccine dose of 1 x 10^5 IU per injection
  Interventions: Biological: AVX101
- Placebo (Placebo Comparator)
  Interventions: Other: placebo

INTERVENTIONS:
Biological: AVX101 — Alphavirus replicon particle vaccine expressing HIV Gag antigen
  Arms: 1 x 10^4 IU dose; 1 x 10^5 IU dose
Other: placebo — phosphate buffered saline, pH 7.2, HSA, sodium gluconate, and sucrose
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if different doses of an experimental HIV vaccine are safe and to study how the immune system responds to the vaccine. The vaccine will be tested in healthy, HIV uninfected volunteers. AVX101 contains only one of the many substances that HIV needs to make more copies of itself; therefore, the vaccine cannot cause HIV or AIDS.

DETAILED DESCRIPTION:
This study was designed to evaluate the safety and immunogenicity of an alphavirus replicon HIV subtype C gag vaccine. This vaccine utilizes a propagation-defective replicon vector system derived from an attenuated strain of Venezuelan Equine Encephalitis (VEE) virus. The vaccine replicon expresses the gag gene from a South African subtype C isolate of HIV-1.

This study evaluated the AVX101 vaccine in healthy, HIV uninfected volunteers in both the United States and South Africa. Participants will be randomized to receive either vaccine or placebo at study entry and again at Months 1 and 3. The study was originally designed to enroll four groups of participants in both the US and South Africa, with successive groups receiving increasing doses of the vaccine, but was later amended to enroll only two groups. Twelve US participants (US Group 1) were randomized to receive either vaccine or placebo. After a review of initial safety data from this group, 12 South African participants (SA Group 1) were randomized to receive the same vaccine dose as US Group 1 or placebo, while 12 US participants (US Group 2) were randomized to receive the next higher vaccine dose or placebo. Review of safety data from SA Group 1 and US Group 2 was used to inform the decision to begin enrollment into SA Group 2 .

Participants had nine study visits over 12 months. Study visits included clinical evaluation, urine and blood tests, and HIV tests. After each injection, participants were asked to record their temperature and any symptoms each day for 7 days and report them to the clinic staff.

ELIGIBILITY:
Inclusion Criteria

* HIV negative
* Willing to receive HIV test results
* Good general health
* Acceptable methods of contraception for females of reproductive potential
* Hepatitis B surface antigen negative
* Anti-hepatitis C virus antibody (anti-HCV) negative or negative HCV PCR if anti-HCV is positive
* Access to participating site and available for follow-up during the 12 month study

Exclusion Criteria

* HIV vaccines or placebos in prior HIV vaccine trial
* Measurable anti-VEE antibody
* High risk for HIV infection according to HVTN Risk Criteria
* Immunosuppressive medications within 168 days prior to first study vaccine administration
* Blood products within 120 days prior to first study vaccine administration
* Immunoglobulin within 60 days prior to first study vaccine administration
* Live attenuated vaccines within 30 days prior to first study vaccine administration
* Investigational research agents within 30 days prior to first study vaccine administration
* Subunit or killed vaccines within 14 days prior to first study vaccine administration
* Current tuberculosis prophylaxis or therapy
* Active syphilis
* Serious adverse reaction to vaccines. A person who had an adverse reaction to pertussis vaccine as a child is not excluded.
* Autoimmune disease or immunodeficiency
* Unstable asthma
* Type 1 or Type 2 Diabetes Mellitus
* Thyroid disease requiring treatment
* Serious angioedema within the past 3 years
* Uncontrolled hypertension
* Bleeding disorder
* Malignancy unless it has been surgically removed and, in the opinion of the investigator, is not likely to recur during the study period
* Seizure disorder requiring medication within the past 3 years
* Asplenia
* Mental illness that would interfere with compliance with the protocol
* Other conditions that, in the judgement of the investigator, would interfere with the study
* Pregnant or breast-feeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2003-07; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Grade IV adverse events | 1 year
  The sample size at each vaccine dose level was selected such that the stopping rule for not escalating the dose (2 or more vaccine-related Grade IV adverse experiences) would be met with high probability if the true toxicity rate was above 15-20%, and such that dose escalation would occur with high probability if the true toxicity rate was less than 5%.

SECONDARY OUTCOMES:
Local and systemic adverse events | 7 days after each dose
  Reactogenicity assessments were performed for all participants before and after each injection, beginning 25 to 45 minutes post injection and continuing daily for 7 days. Assessments performed included systemic reactogenicity (body temperature, malaise and/or fatigue, myalgia, headache, chills, arthralgia, nausea, vomiting) and local reactogenicity (injection site pain, tenderness, erythema or induration, and axillary lymph node tenderness or enlargement).
Binding antibodies by ELISA | 1 year
  Binding antibodies to commercially available Gag protein (P55 Gag; Quality Biologicals) were assessed by ELISA using single serum dilutions (1/50 or 1/100) on samples taken at baseline, two weeks after the second and third vaccinations and at the final visit. Samples that were positive in the initial ELISA were tested by endpoint titration ELISA using six 2- to 7-fold serial dilutions of serum beginning at a 1/50 or 1/100 dilution. Magnitude of responses is reported as the difference in optical density (OD) in antigen-containing and non-antigen containing wells at the 1:50 dilution.
Chromium release CTL assay | 3 months
  A standard 51Cr-release CTL assay was performed on fresh peripheral blood mononuclear cells (PBMC) at baseline and 2 weeks after the second and third vaccinations, using a 50:1 effector to target (E:T) ratio.
IFN-gamma ELISpot assay | 3 months
  Bulk T cell responses were assessed by IFN-γ ELISpot, using cryopreserved PBMC collected at baseline and 2 weeks after the second and third vaccinations, and stimulated overnight with Gag peptide pools at 200,000 cells per well.
Antibodies to VEE virus | 1 year
  Neutralizing antibodies to VEE virus were measured in serum obtained at baseline, 2 weeks after the second and third vaccinations and at the final visit.
Replication-competent viral vector viremia | 2 weeks after each vaccine dose
  Any participant who reported a fever greater than 38oC, or other moderate symptoms consistent with a viral illness (e.g. headache or malaise) during the 7 days following vaccination, or neurological symptoms (e.g. nuchal rigidity, ataxia, convulsions, coma, paralysis) within the window of the 2-week post vaccination visit, provided a serum sample to confirm the absence of replication-competent VEE viremia.
Lymphoproliferation assay | 1 year
  A lymphocyte proliferation assay in response to purified Gag protein and/or Gag peptides was performed on cryopreserved PBMC collected at baseline, 2 weeks after the second and third vaccinations, and at the final visit.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Burke, MD, Study Chair — Johns Hopkins University; Salim Abdool Karim, MD, PhD, Study Chair — University of Natal, Durban, South Africa
Locations (7):
- United States (5):
  - Johns Hopkins University, Baltimore, Maryland
  - Columbia University, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - New York Blood Ctr- Union Square, The Bronx, New York
  - Vanderbilt University, Nashville, Tennessee
- South Africa (2):
  - SAAVI Vaccine Research Unit, Durban
  - Chris Hani Baragwanath Hospital, Soweto

REFERENCES:
- [Background] Pushko P, Parker M, Ludwig GV, Davis NL, Johnston RE, Smith JF. Replicon-helper systems from attenuated Venezuelan equine encephalitis virus: expression of heterologous genes in vitro and immunization against heterologous pathogens in vivo. Virology. 1997 Dec 22;239(2):389-401. doi: 10.1006/viro.1997.8878. PMID 9434729
- [Background] Pushko P, Bray M, Ludwig GV, Parker M, Schmaljohn A, Sanchez A, Jahrling PB, Smith JF. Recombinant RNA replicons derived from attenuated Venezuelan equine encephalitis virus protect guinea pigs and mice from Ebola hemorrhagic fever virus. Vaccine. 2000 Aug 15;19(1):142-53. doi: 10.1016/s0264-410x(00)00113-4. PMID 10924796
- [Background] Davis NL, Caley IJ, Brown KW, Betts MR, Irlbeck DM, McGrath KM, Connell MJ, Montefiori DC, Frelinger JA, Swanstrom R, Johnson PR, Johnston RE. Vaccination of macaques against pathogenic simian immunodeficiency virus with Venezuelan equine encephalitis virus replicon particles. J Virol. 2000 Jan;74(1):371-8. doi: 10.1128/jvi.74.1.371-378.2000. PMID 10590126
- [Background] Strauss JH, Strauss EG. The alphaviruses: gene expression, replication, and evolution. Microbiol Rev. 1994 Sep;58(3):491-562. doi: 10.1128/mr.58.3.491-562.1994. PMID 7968923
- [Derived] Wecker M, Gilbert P, Russell N, Hural J, Allen M, Pensiero M, Chulay J, Chiu YL, Abdool Karim SS, Burke DS; HVTN 040/059 Protocol Team; NIAID HIV Vaccine Trials Network. Phase I safety and immunogenicity evaluations of an alphavirus replicon HIV-1 subtype C gag vaccine in healthy HIV-1-uninfected adults. Clin Vaccine Immunol. 2012 Oct;19(10):1651-60. doi: 10.1128/CVI.00258-12. Epub 2012 Aug 22. PMID 22914365